CLINICAL TRIAL: NCT06164587
Title: A Non-Randomized, Open Label, Safety and Efficacy Study Evaluating Kamuvudine-8 (K8) for the Treatment of Patients With Geographic Atrophy
Brief Title: Evaluation of Kamuvudine-8 in Subjects With Geographic Atrophy
Acronym: K8 for GA
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Michelle Abou-Jaoude (Other)
Collaborators: Inflammasome Therapeutics (Industry)
Responsible Party: Sponsor-Investigator, Michelle Abou-Jaoude, Assistant Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 91507
Record Dates: First submitted 2023-12-01; First posted 2023-12-11 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Geographic Atrophy; Age-Related Macular Degeneration
Keywords: ophthalmology; K8; kamuvudine
MeSH Terms: conditions — Geographic Atrophy; Macular Degeneration | interventions — Potassium, Dietary

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Patients with geographic atrophy associated with age-related macular degeneration (Experimental): Kamuvudine-8 treatment (0.3 mg) at baseline visit and week 13 visit, in one eye of each subject, for a total of up to 30 subjects. When new study drug is received, the next 20 patients will be enrolled to receive K8 treatment (either 0.7 mg or 1.05 mg) at baseline and week 13, in one eye of each subject, for a total of up to 30 subjects. The total of 30 patients is across three dosing groups. Once subjects have received one dose/type of implant, there is no crossover to a different group.
  Patients will be followed for 26 weeks after baseline visit injection.
  Interventions: Drug: K8

INTERVENTIONS:
Drug: K8 — sustained released bio-erodible intravitreal implants
  Other Names: SOM-401

SUMMARY:
This interventional study is a single-center, open label, 26-week study, designed to evaluate the safety and treatment efficacy of K8 in patients with geographic atrophy (GA) due to age-related macular degeneration (AMD). Up to 5 subjects will receive study medication. Study treatment will be administered by intravitreal injections. Number of participants has been expanded to 30.

Participants will have 7 scheduled visits - Screening with baseline (injection), safety visit 2 days after injection, week 4, week 13 (injection), safety visit 2 days after injection, week 17, week 26.

Exams will look for continuous changes in visual acuity, change in area of geographic atrophy lesions in diagnostic imaging, response measured by multifocal electroretinogram, change in reading speed, and change in microperimetry response.

ELIGIBILITY:
Inclusion Criteria:

* Aged 50 or older, diagnosed with geographic atrophy (GA) due to age-related macular degeneration (AMD).
* Best corrected visual acuity (BCVA) 24 or greater Early Treatment of Diabetic Retinopathy Study (ETDRS) letters (approximately Snellen 20/320 or greater), in study eye.
* The entire geographic atrophy (GA) lesion must be completely visualized on the macula centered image and must be able to be imaged in its entirety and not contiguous with any areas of peripapillary atrophy except in such cases where there is a "neck" or some narrow area connecting the GA with the peripapillary atrophy, as determined by Fundus Autofluorescence (FAF) imaging at screening:
* Both eyes must have GA and the total GA area in each eye must be ≥ 2.5 and ≤ 20.0 mm2 (1 and 8 disk areas [DA] respectively)
* If geographic atrophy (GA) is multifocal, at least one focal lesion must be ≥ 1.25 mm2 (0.5 DA), with the overall aggregate area of GA, as specified above.
* If geographic atrophy (GA) is unifocal, then the lesion must be extrafoveal.
* Presence of any pattern of hyperautofluorescence in the junctional zone of geographic atrophy (GA). Absence of hyperautofluorescence (i.e., pattern = none) is exclusionary.
* Fundus Autofluorescence (FAF), spectral-domain optical coherence tomography (SD-OCT), or Fluorescein Angiography (FA) imaging of entire geographic atrophy (GA)lesion at least 6 months prior to entry.

General Exclusion Criteria:

* Females who are pregnant, nursing, planning a pregnancy or who are of childbearing potential not using a reliable method of contraception
* History or current evidence of hypersensitivity to any components of the study medication or fluorescein, as assessed by the investigator
* Participation in any investigational drug or device study within 30 days prior to baseline
* History or current evidence of a medical condition or medication use that may, in the opinion of the investigator, preclude the safe administration of study medication or affect the results of the study
* Participation in any systemic experimental treatment or any other systemic investigational new drug within 6 weeks or 5 half-lives of the active ingredient (whichever is longer) prior to the start of study treatment. Clinical trials solely involving observation, over-the-counter vitamins, supplements, or diets are not exclusionary.

Ocular Exclusion Criteria:

* Active ocular or periocular infections, malignancy
* History of major ophthalmic surgery in the past 3 months, and any ophthalmic surgery in study eye in the last 30 days
* History of significant ocular disease other than AMD that may confound results
* Any history or current evidence of exudative ("wet") AMD including any evidence of retinal pigment epithelium rips or evidence of retinal, choroidal, or peripapillary neovascularization in either eye
* Known hypersensitivity to study drug or any of the excipients in implant
* Macular atrophy secondary to a condition other than AMD
* History of laser therapy in the macular region
* Aphakia or surgically compromised/absent posterior capsule including presence of scleral fixated lenses. Note: YAG laser posterior capsulotomy for posterior capsule opacification done at least 60 days prior to screening is not exclusionary
* History of prior posterior vitrectomy
* History of prior intraocular gene therapy for any indication
* History of extended hydroxychloroquine or pentosan polysulfate exposure (> 3 months)
* Current use of medications known to be toxic to the lens, retina, or optic nerve (e.g., deferoxamine, chloroquine/hydroxychloroquine [Plaquenil®], tamoxifen, phenothiazines, ethambutol, digoxin, pentosan polysulfate, and aminoglycosides).
* Uncontrolled glaucoma (defined as intraocular pressure >21mm Hg despite treatment with ocular hypotensive medications at baseline)
* Prior participation in another interventional clinical study or treatment for GA in the study eye including topical, IVT, subretinal, suprachoroidal, periocular or oral medication or placebo within 5 half-lives of the active ingredient

Prohibited Medications/Treatments:

* Systemic anti-VEGF medications
* Intravitreal injections of Syfovre (pegcetacoplan), Izervay (avacincaptad pegol) or other complement inhibitors in either eye
* Gene therapy injections in either eye

Ages: 50 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-04-18 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Adverse Events | Within the study period (of 26 weeks)
  Frequency of participants experiencing ocular or systemic adverse events.
Mean change in best-corrected visual acuity (BCVA) | At baseline visit, week 13 visit, and week 26 visit
  best-corrected visual acuity as defined by the number of letters read on the scale set by the ETDRS (Early Treatment of Diabetic Retinopathy Study). (More letters read equates to better visual acuity)
Mean change in low-luminance best-corrected visual acuity (ll-BCVA) | At baseline visit, week 13 visit, and week 26 visit
  best-corrected visual acuity in low-lighting settings
Change in size of geographic atrophy (GA) on fundus autofluorescence (FAF) | At baseline visit, week 13 visit, and week 26 visit
  Change in total area of geographic atrophy lesions as analyzed with FAF imaging over the course of the trial
change in size of geographic atrophy (GA) on optical coherence tomography (OCT) | At baseline visit, week 13 visit, and week 26 visit
  Change in total area of geographic atrophy lesions as analyzed with OCT imaging
change in size of geographic atrophy (GA) on fluorescein angiogram (FA) | At baseline visit, week 13 visit, and week 26 visit
  Change in total area of geographic atrophy lesions as analyzed with FA imaging
Change in multifocal electroretinograms (mfERG) response | At baseline visit, week 13 visit, and week 26 visit
  Total response change measured by mfERG (performed upon site PI discretion and only if site has), which measures the electrical signal generated by a functionining eye processing information
Change in microperimetry response | At baseline visit, week 13 visit, and week 26 visit
  change in response to visual field testing with microperimetry (undilated) over the course of the study (performed upon site PI discretion and only if site has).
Change in reading speed | At baseline visit, week 13 visit, and week 26 visit
  Change in reading speed as measured by Radner reading chart procedure
Discontinued subjects | This will be done at every scheduled visit and any unscheduled visit, as well as when reported by participants (for 26 weeks)
  Number of subjects exiting study for any reason

SECONDARY OUTCOMES:
Change in best corrected visual acuity (BCVA) over multiple time points | Day 2 visit, Week 4 visit, Week 13 visit, Week 13 + 2 Days visit, and Week 17 visit
  Change in best corrected visual acuity (BCVA) at each study visit

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Abou-Jaoude, MD, Principal Investigator — University of Kentucky
Locations (9):
- United States (9):
  - Loma Linda University, Loma Linda, California
  - University of Kentucky Advanced Eye Care, Lexington, Kentucky
  - The Maine Eye Center, Portland, Maine
  - Oregon Eye Consultants, Cascade Medical Research, Eugene, Oregon
  - Hilton Head Retina Institute, Hilton Head, South Carolina
  - Ophthalmology LTD, Sioux Falls, South Dakota
  - Southeastern Retina Associates, Hixson, Tennessee
  - Southeastern Retina Associates, Bristol, Virginia
  - Vistar Eye Center, Roanoke, Virginia

IPD SHARING:
Plan to Share IPD: No